CLINICAL TRIAL: NCT05686876
Title: Fibroblast Activation Protein-Targeted PET/CT With 68Ga-FAPI for Imaging Psoriatic Arthritis: Comparison to 18F-NAF PET/CT
Brief Title: FAPI-PET/CT in Psoriatic Arthritis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: LXM-230107
Record Dates: First submitted 2023-01-07; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — 68Ga-FAPI

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI, PET/CT (Experimental): Inject 68Ga-FAPI and then perform PET/CT scan.
  Interventions: Drug: 68Ga-FAPI

INTERVENTIONS:
Drug: 68Ga-FAPI — Intravenous injection of one dosage of 74-148 MBq (2-4 mCi) 68Ga-FAPI. Tracer doses of 68Ga-FAPI will be used to image lesions of PsA by PET/CT.
  Other Names: 68Ga-fibroblast activating protein inhibitors

SUMMARY:
68Ga-FAPI has been developed as a tumor-targeting agent as fibroblast activation protein is overexpressed in cancer-associated fibroblasts and some inflammation, such as IgG4-related disease. Therefore, this prospective study is going to investigate whether 68Ga-FAPI PET/CT may be superior for disease activity assessment and follow-up of psoriatic arthritis than 18F-NAF PET/CT.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is a chronic inflammatory disease that develops in up to 30% of patients with psoriasis and characterized by diverse clinical features including peripheral and axial arthritis, enthesitis, dactylitis and nail dystrophy, leading to impaired function and reduced quality of life. Positron emission tomography (PET) allows for highly sensitive depiction of targets at the molecular level and can be used to specifically visualize immune cells of interest through the use of specific tracers. In this study, we used two tracers: 68Ga-fibroblast activation protein inhibitor (FAPI) and 18F-sodium fluoride (18F-NaF) to evaluate both joint inflammation and bone metabolism in patients with PsA. And the study is going to investigate whether 68Ga-FAPI PET/CT may be superior for disease activity assessment and follow-up of psoriatic arthritis than 18F-NAF PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* fulfilled the 2006 Classification Criteria for Psoriatic Arthritis (CASPAR)
* 18F-NAF PET/CT within two weeks
* signed written consent.

Exclusion Criteria:

* pregnancy
* breast feeding
* known allergy against FAPI
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | Through study completion, an average of 3months
  Diagnostic value of 68Ga-FAPI PET/CT for PsA in comparison with 18F-FDG PET/CT.

SECONDARY OUTCOMES:
Disease activity assessment | Through study completion, an average of 3months.
  Correlation between disease activity assessed on 68Ga-FAPI PET/CT and clinical parameters for PsA.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Yang F, Lu C, Pan Q, Zhang R, Yang M, Wang Q, Li M, Zeng X, Luo Y, Leng X. 68Ga-FAPI and 18F-NaF PET/CT in psoriatic arthritis: a comparative study. Rheumatology (Oxford). 2025 May 1;64(5):2575-2582. doi: 10.1093/rheumatology/keae577. PMID 39576694